CLINICAL TRIAL: NCT01147380
Title: A Novel Immunotherapy for Liver Transplant Patients With Hepatocellular Carcinoma: Anti-tumor Effect of IL2-activated Donor Liver Natural Killer Cell
Brief Title: Safety Study of Liver Natural Killer Cell Therapy for Hepatoma Liver Transplantation
Acronym: MIAMINK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seigo Nishida (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Sponsor-Investigator, Seigo Nishida, Professor of clinical surgery, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20100344; 20100344 (Other: University of Miami IRB number)
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Liver Cirrhosis; Hepatocellular Carcinoma; Evidence of Liver Transplantation
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Small dose (Experimental): From the donor liver perfusate, mononuclear cell will be extracted and cultured. Then, the cells will be stimulated with IL-2. The number of inoculation cells( mainly NK cells) is between 10 and 100 million cells. The cells will be given to the liver transplant recipient who had the same donor for liver and liver perfusate. Patient of this arm receive small dose of liver NK cell inoculation as described.
  Interventions: Biological: Liver NK cell inoculation
- Large dose (Experimental): From the donor liver perfusate, mononuclear cell will be extracted and cultured. Then, the cells will be stimulated with IL-2. The number of inoculation cells(mainly NK cells) is between 100 and 1000 million cells. The cells will be given to the liver transplant recipient who had the same donor for liver and liver perfusate.Patient of this arm receive large dose of liver NK cell inoculation as described.
  Interventions: Biological: Liver NK cell inoculation

INTERVENTIONS:
Biological: Liver NK cell inoculation — Liver transplant recipients will receive once liver NK cell inoculation several days after liver transplantation.

SUMMARY:
The objective of this study is to evaluate feasibility and safety of the adoptive transfer of activated natural killer (NK) cells extracted from cadaveric donor liver graft perfusate for liver transplant recipients with hepatocellular carcinoma (HCC)

DETAILED DESCRIPTION:
To investigate whether adoptive transfer of IL-2 stimulated NKcells extracted from cadaveric donor liver graft exudates into recipient with HCC will lead to prevent recurrence of HCC after liver transplantation.

The method we plan to use is to collect NK cells from the cadaveric donor liver perfusate at the time of organ recovery. The perfusate will be condensed by centrifuging and liver mononuclear cells (LMNC) were isolated by gradient centrifugation. LMNC will be cultured with anti-CD3 antibody. LMNC will be separted into a CD3-/CD56+ NK cell fraction and a non-NK cell fraction. The purity of isolated fractions will be assessed by Flow cytometric analyses. NK cells will be cultured with human recombinant IL-2 in 10% RPMI at 37 ºC in a 5% CO2 incubator. NK cells will be infused intravenously to the recipient with HCC who have liver transplant from the same cadaveric donor at post operative day 4 in attempt to prevent the metastasis and recurrence of HCC.

ELIGIBILITY:
Inclusion Criteria:

* Primary liver transplant recipient with HCC
* Patients need to meet the liver transplant eligibility criteria
* Cardiac function; cardiac echo will indicate that ejection fraction (EF) > 35% or right ventricular systolic pressure (RVSP) < 50mmHg. Stress echo will show no ischemic lesion (if applicable).
* Pulmonary function; SpO2 >90% or PaO2 > 60 mmHg, or CT will show no active pulmonary lesion.
* Complete blood count; Platelet > 20,000 /mm^3, Hematocrit > 20%, WBC > 1,000 /mm^3
* Eighteen years of age or older
* Ability to provide informed consent
* If female of childbearing potential:

Must not be lactating, must have a negative serum B-human chorionic gonadotropin (HCG) test within 7 days prior to Day of Transplant, and must agree to practice an acceptable and reliable form of contraception during the study Ability to provide informed consent

Exclusion Criteria:

* Living donor liver transplant; a healthy person donates part of his or her liver to the recipient
* Multiple organ transplants
* Prior solid organ or bone marrow transplant recipients
* Fluminant hepatic failure
* The patients regularly receive the hemodialysis more than twice a week before liver transplant
* Status 1 transplants; acute severe disease and defined as a patient with only recent development of liver disease who is in the intensive care unit of the hospital with a life expectancy without a liver transplant of fewer than 7 days
* ABO incompatible transplants
* Transplants utilizing livers from non-heart beating donors; the cardiac death donor
* Recipients of investigational therapy within 90 days prior to transplant procedure
* Acute viral illness
* History of malignancy within 5 years, with exception of: Adequately treated localized squamous or basal cell carcinoma of the skin without evidence or recurrence, and/or Hepatocellular carcinoma
* Illness other than primary liver disease (e.g., severe ischemic heart disease, left ventricular dysfunction, or pulmonary disease), which, in the opinion of the Investigator, may significantly increase the risk of the transplantation procedure
* Current drug or alcohol abuse or, in the opinion of the Investigator, is at risk for poor compliance (no drug testing required)
* Serology positive donor (HCV, HBsAg, HBcAb, HTLV-1, HTLV-3, EBVIgM)
* Poor liver function donor (Total bilirubin > 3.0 mg/dl, Prothrombin time > 35 sec),
* Patients who receive intercurrent chemotherapy at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seigo Nishida, MD PhD, Principal Investigator — Department of Surgery, University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ohira M, Hotta R, Tanaka Y, Matsuura T, Tekin A, Selvaggi G, Vianna R, Ricordi C, Ruiz P, Nishida S, Tzakis AG, Ohdan H. Pilot study to determine the safety and feasibility of deceased donor liver natural killer cell infusion to liver transplant recipients with hepatocellular carcinoma. Cancer Immunol Immunother. 2022 Mar;71(3):589-599. doi: 10.1007/s00262-021-03005-3. Epub 2021 Jul 19. PMID 34282496

RESULTS

PARTICIPANT FLOW:
Groups:
- Small Dose: The number of inoculation cells is between 10 and 100 million cells.
  Liver NK cell inoculation: Liver transplant recipients will receive liver NK cell inoculation several days after liver transplantation.
- Large Dose: The number of inoculation cells is between 100 and 1000 million cells
  Liver NK cell inoculation: Liver transplant recipients will receive liver NK cell inoculation several days after liver transplantation.
Period: Overall Study
Arm/Group | Small Dose | Large Dose
Started | 6 | 12
Completed | 6 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Small Dose: The number of inoculation cells is between 10 and 100 million cells.
  Liver NK cell inoculation: Liver transplant recipients will receive once liver NK cell inoculation several days after liver transplantation.
- Large Dose: The number of inoculation cells is between 100 and 1000 million cells
  Liver NK cell inoculation: Liver transplant recipients will receive once liver NK cell inoculation several days after liver transplantation.
- Total: Total of all reporting groups
Arm/Group | Small Dose | Large Dose | Total
Number analyzed (Participants) | 6 | 12 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 10 | 15
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: years] | 59.5 [52 to 66] | 55.6 [20 to 68] | 56.9 [20 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 6 | 10 | 16
Region of Enrollment [Number; unit: participants]
  United States | 6 | 12 | 18

OUTCOME MEASURES:

1. Primary Outcome: Side Effect of Cadaveric Donor Liver NK Cell Infusion
Description: Side effect of cadaveric donor liver NK cell infusion We will measure the occurence of the side effect of the liver NK cell infusion. We will monitor the patient condition clinically. If any side effect are noticed, we will record them and report to the data safety monitoring comittee.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Small Dose | Large Dose
Number analyzed (Participants) | 6 | 12
participants | 0 | 0

2. Secondary Outcome: NK Cell Infusion-related Toxicity
Description: To assess NK cell infusion -related toxicity at the bedside. We will monitor the patient and check the vital sign. If any side effect are noticed, we will record and report to the data safety monitoring comittee.
Time Frame: 1 year
Population: Participants were devided two group( small and large dose) as described based on the dose of infused cell numbers.
Measure: Number; unit: participants
Arm/Group | Small Dose | Large Dose
Number analyzed (Participants) | 6 | 12
participants | 0 | 0

3. Secondary Outcome: Anti-HCC Effect of This Treatment
Time Frame: 2 year
Reporting Status: Not Posted

4. Secondary Outcome: Anti-HCV Effect of This Treatment (If Applicable)
Time Frame: 2 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events will be graded according to the Common terminology criteria for Adverse Events Guide.
  A Data Safety Monitoring Committee will be constituted to analyze safety and preliminary evidence of efficacy of the trial.
  Adverse events will be reported to the IRB and DSMB. Serious adverse events will be reported to the DSMB within 24 hours.
Arm/Group | Small Dose | Large Dose
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 0/6 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Small Dose (N=6) | Large Dose (N=12)
fatigue (General disorders) | 0 (0) | 0 (0) — General fatigue and tiredness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes